CLINICAL TRIAL: NCT04950257
Title: Evaluating the Effects of a Self-help Mobile Phone Application on Worry and Rumination Experienced by Young Adults: a Preventative Intervention for Depression and Anxiety
Brief Title: Evaluating the Effects of a Self-help Mobile Phone Application on Worry and Overthinking in Young Adults Aged Between 16 and 24.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Principal Investigator, Daniel Edge, Trainee Clinical Psychologist, University of Exeter
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: eCLESPsy001977
Record Dates: First submitted 2021-06-22; First posted 2021-07-06 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Rumination; Worry; Repetitive Negative Thinking
MeSH Terms: conditions — Rumination Syndrome

STUDY DESIGN:
Intervention Model Description: The trial design is of a superiority two-arm parallel-group single-blind randomised controlled trial comparing usual practice plus up to 6 weeks of using the repetitive negative thinking-targeting digital self-help app versus usual practice and waiting list control. The primary hypothesis is that the rumination-targeting digital self-help app will reduce rumination and worry significantly more than waiting list control at 6 weeks follow-up.
Who Masked: Outcomes Assessor
Masking Description: The analysis team members will be blind to the randomisation process and group allocation of participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- waiting list control group (Active Comparator): Participants randomly allocated to this arm will be offered self-help components within a mobile phone app to target worry and rumination after a 6-week wait.
  Interventions: Device: digital CBT self-help including specific intervention elements to target worry and rumination.
- treatment group (Experimental): Participants randomly allocated to this arm will be offered self-help components within a mobile phone app to target worry and rumination immediately.
  Interventions: Device: digital CBT self-help including specific intervention elements to target worry and rumination.

INTERVENTIONS:
Device: digital CBT self-help including specific intervention elements to target worry and rumination. — The self-help app includes self-monitoring, psychoeducation and active self-help exercises. The self-monitoring includes daily mood ratings and an ecological momentary assessment option (MoodTracker) for more detailed analysis of mood, worry, activity and situational context. The digital self-help provides psychoeducation, tips, advice, exercises and training for each individual focused on reducing worry and rumination, using strategies from the proven rumination-focused CBT intervention. The app includes text, pictures, audio-recordings, animations, audio-exercises to practice (e.g., self-compassion, relaxation, concreteness exercises), and questionnaires with tailored feedback. The app is designed for iOS and Android use.
  Other Names: MyMoodCoach

SUMMARY:
This project seeks to understand if a new self-help mobile phone application (called MyMoodCoach) is effective at reducing worry and overthinking, prominent risk factors that predict reduced well-being and poor mental health. As a primary outcome, the investigators are predicting that people who use the app will report more significant reductions on measures of overthinking than those who do not. The investigators also predict that people who use the app will report more significant reductions in measures of worry as well as reported symptoms of depression and anxiety. Further, it is predicted that people who use the app will report a significantly higher increase in their well-being compared to those who do not.

DETAILED DESCRIPTION:
The Emotional Competence for Well-Being in Young Adults study has developed an emotional competence app to be examined via cohort multiple randomised controlled trial (cmRCT) in a longitudinal prospective cohort. This off-shoot study adapts the app to focus on targeting worry and overthinking (also known as rumination), which are prominent risk factors for poor mental health.

Within this study, 16-24-year-olds in the UK, who report elevated worry and rumination on standardised questionnaires are randomised to either receive the mobile phone app immediately or to receive the app after a wait of 6 weeks. In total, the study will aim to recruit 204 participants across the UK. Assessments take place at baseline (pre-randomisation), 6 and 12 weeks post-randomisation. Primary endpoint for the study is the change in levels of rumination assessed at 6 weeks after randomisation. Worry, depressive symptoms, anxiety symptoms and well-being are secondary outcomes. Compliance, adverse events, and potentially mediating variables will be carefully monitored.

This trial aims to provide a better understanding of the benefits of tackling rumination and worry via an intervention delivered via mobile phone app with respect to promoting well-being and preventing poor mental health in young people. This prevention mechanism trial will establish whether targeting worry and rumination directly via an app provides a feasible approach to prevent depression and anxiety, with scope to become a widescale public health strategy for preventing poor mental health and promoting well-being in young people.

ELIGIBILITY:
Inclusion Criteria:

* aged 16 to 24 years old (inclusive)
* currently based in the UK
* possess a basic literacy in English
* able to provide informed consent
* reporting elevated levels of worry and rumination, defined here as scoring above the 50th percentile (i.e., top-half of scale) on either the RSS (>34) or the PSWQ (>41)
* have regular access to a smartphone (android or iOS).

Exclusion Criteria:

* reporting highly elevated symptoms of depression indicating more specialist treatment is required (PHQ-9 > 20)
* self-report of active suicidality
* self-report currently receiving psychological therapy, counseling, or psychiatric medication, including antidepressants, for a current mental health condition

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 236 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Change in rumination using the Ruminative Response Scale (RRS) | Change from baseline at 6 weeks
  A well established 22-item measure of pathological rumination which predicts subsequent depression.

SECONDARY OUTCOMES:
Change in worry using the Penn State Worry Questionnaire (PSWQ) | Change from baseline at 6 weeks
  a well-validated 16-item measure of trait tendency towards worry
Change in symptoms for depression using the Patient Health Questionnaire-9 (PHQ-9) | Change from baseline at 6 weeks
  a well-validated measure of depression and depressive symptoms
Change in wellbeing using the Warwick-Edinburgh Mental Well Being Scale (WEMWBS) | Change from baseline at 6 weeks
  a leading validated self-reported index of well-being with excellent psychometric properties comprising 14 items
Change in symptoms for anxiety using the Generalized Anxiety Disorder-7 (GAD-7) | Change from baseline at 6 weeks
  A well validated measure of anxiety and anxiety symptoms

OTHER OUTCOMES:
Change in worry using the Penn State Worry Questionnaire (PSWQ) | Change from 6 weeks post randomisation at 12 weeks post randomisation
  a well-validated 16-item measure of trait tendency towards worry
Change in rumination using the Ruminative Response Scale (RRS) | Change from 6 weeks post randomisation at 12 weeks post randomisation
  A well established 22-item measure of pathological rumination which predicts subsequent depression.
Change in symptoms for depression using the Patient Health Questionnaire-9 (PHQ-9) | Change from 6 weeks post randomisation at 12 weeks post randomisation
  a well-validated measure of depression and depressive symptoms
Change in wellbeing using the Warwick-Edinburgh Mental Well Being Scale (WEMWBS) | Change from 6 weeks post randomisation at 12 weeks post randomisation
  a leading validated self-reported index of well-being with excellent psychometric properties comprising 14 items
Change in symptoms for anxiety using the Generalized Anxiety Disorder-7 (GAD-7) | Change from 6 weeks post randomisation at 12 weeks post randomisation
  A well validated measure of anxiety and anxiety symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ed R Watkins, Professor, Study Director — Exeter University; Dan J Edge, MRes, Principal Investigator — Exeter University
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant and clinical and economic data reported in publications will be made available through the University of Exeter's Institutional Repository - Open Research Exeter (see https://ore.exeter.ac.uk).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol and informed consent form will be uploaded with this registration. The SAP is included in the study protocol.
  Data Access: Post-analysis, the final anonymised dataset will preferentially be stored in Open Research Exeter (ORE), the University of Exeter's open access repository. The data will be available from 24 months after trial completion (end of December 2021).
Access Criteria: Access to these data is permitted but controlled through requests made via the repository to a review panel from the trial team, led by the chief investigator, which will assess requests on scientific merit and commercial sensitivity. Although use is permitted, this will be on the basis that the source of the data is acknowledged (including the funder) and it includes reference to the data set 'handle', and a data access agreement is signed, subject to approval by funder.

REFERENCES:
- [Background] Edge D, Newbold A, Ehring T, Rosenkranz T, Frost M, Watkins ER. Reducing worry and rumination in young adults via a mobile phone app: study protocol of the ECoWeB (Emotional Competence for Well-Being in Young Adults) randomised controlled trial focused on repetitive negative thinking. BMC Psychiatry. 2021 Oct 21;21(1):519. doi: 10.1186/s12888-021-03536-0. PMID 34674669
- [Derived] Edge D, Watkins E, Newbold A, Ehring T, Frost M, Rosenkranz T. Evaluating the Effects of a Self-Help Mobile Phone App on Worry and Rumination Experienced by Young Adults: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2024 Aug 13;12:e51932. doi: 10.2196/51932. PMID 39137411